CLINICAL TRIAL: NCT00833495
Title: A Multi-Center, Randomized, Double-Masked Evaluation of the Efficacy of Co-Administration of FOV1101-00 (Cyclosporine 0.01% or 0.02%) and Prednisolone Acetate 0.12% (PredMild®) Compared to Prednisolone Acetate 1% Alone or Vehicle Alone in Patients With Mild Ongoing Ocular Allergic Inflammation
Brief Title: Evaluation of Efficacy of Coadministration of FOV1101-00 and Prednisolone Acetate in Patients With Mild Ongoing Ocular Allergic Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fovea Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 08-003-27
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): FOV1101-00 concentration 1 and Prednisolone Acetate 0.12% (Pred Mild®)
  Interventions: Drug: Prednisolone Acetate 0.12% (Pred Mild®); Drug: FOV1101-00
- 2 (Experimental): FOV1101-00 concentration 2 and Prednisolone Acetate 0.12% (Pred Mild®)
  Interventions: Drug: Prednisolone Acetate 0.12% (Pred Mild®); Drug: FOV1101-00
- 3 (Experimental): Vehicle of FOV1101-00 and Prednisolone Acetate 1% (Pred Forte®)
  Interventions: Drug: Prednisolone Acetate 1% (Pred Forte®); Drug: Placebo
- 4 (Placebo Comparator): Vehicle of FOV1101-00 and vehicle of FOV1101-00
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone Acetate 0.12% (Pred Mild®) — Indicated for the treatment of mild to moderate noninfectious allergic and inflammatory disorders of the lid, conjunctiva, cornea, and sclera (including chemical and thermal burns). Instill one to two drops into the conjunctival sac two to four times daily. During the initial 24 to 48 hours, the dosing frequency may be increased if necessary.
  Arms: 1; 2
Drug: FOV1101-00 — This investigational drug is a low dose cyclosporine (also known as cyclosporine A; CsA) formulation for topical ocular administration. FOV1101-00 is presented as a solution for topical ophthalmic administration in two strengths, concentration 1 or concentration 2 w/v cyclosporine in citrate buffered aqueous vehicle. Application is intended as four times per day.
  Arms: 1; 2
Drug: Prednisolone Acetate 1% (Pred Forte®) — PRED FORTE® is indicated for the treatment of steroid-responsive inflammation of the palpebral and bulbar conjunctiva, cornea, and anterior segment of the globe. Instill one to two drops into the conjunctival sac two to four times daily. During the initial 24 to 48 hours, the dosing frequency may be increased if necessary. Care should be taken not to discontinue therapy prematurely.
  Arms: 3
Drug: Placebo — The vehicle is an eye drop that contains only the inactive ingredients of FOV1101-00.
  Arms: 3; 4

SUMMARY:
This is a phase 2 study that will consist of 3 visits during a 3 week period conducted at up to 5 sites. The purpose of this study is to determine how effective the combination of Pred Mild® and FOV1101-00 is compared to either Pred Forte® alone or to vehicle alone in the prevention of eye allergies. Study subjects will be randomized to one of the following:

* FOV1101-00 concentration 1 and Pred Mild®
* FOV1101-00 concentration 2 and Pred Mild®
* Vehicle of FOV1101-00 and Pred Forte®
* Vehicle of FOV1101-00 and Vehicle of FOV1101-00

ELIGIBILITY:
Inclusion Criteria:

* history of ocular allergies and a positive skin test reaction to allergens within the past 24 months and a history of chronic eye irritation;

Exclusion Criteria:

* active ocular infection; clinically significant blepharitis; follicular conjunctivitis; iritis; any type of glaucoma; ocular surgery within past 3 months; pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Ocular Allergic signs and symptoms Diary Scores | Between V2 and V3

SECONDARY OUTCOMES:
Various ocular and nasal allergic diary scores | Between V2 and V3

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Combal, PharmD, Study Director — Fovea Pharmaceuticals SA
Locations (1):
- Ora, Andover, Massachusetts, United States